CLINICAL TRIAL: NCT00374725
Title: Treatment of Ulcerative Colitis With a Combination of Lactobacillus Rhamnosus and Lactobacillus Acidophilus. A Randomised Placebo Controlled Trial
Brief Title: Treatment of Ulcerative Colitis With a Combination of Lactobacillus Rhamnosus and Lactobacillus Acidophilus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other); Crohn's and Colitis Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VF 20020197
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Last update posted 2006-09-11 (Estimated); Status verified 2002-11

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; Probiotic; Placebo controlled trial; Lactobacillus rhamnosus; Lactobacillus acidophilus
MeSH Terms: conditions — Colitis, Ulcerative

INTERVENTIONS:
Behavioral: Administration of probiotic (L. rhamnosus and L. acidophilus)

SUMMARY:
In this trial we test the hypothesis that a probiotic containing Lactobacillus acidophilus and Lactobacillus rhamnosus is an effective therapy for patients with ulcerative colitis.

DETAILED DESCRIPTION:
In the recent years there has been an increasing interest in the relationship between the gastrointestinal flora and gut function. Several studies have shown promising results for the use of probiotics in patient with inflammatory bowel disease.

In this trial approximately 100 patients with ulcerative colitis will receive treatment with probiotic or placebo for 8 to 10 months as adjuvant therapy.

The trial is double-blind, randomised and controlled.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known ulcerative colitis
* At least one prior flare of the disease
* Clinically and endoscopically active disease
* Age: 18 and above

Exclusion Criteria:

* Changes in azathioprine dosage within the last three months
* Patients with toxic megacolon, peritoneal reaction or severe colonic bleeding
* Known immunodeficiencies
* On-going infectious disease
* On-going treatment with NSAID or cholestyramine
* Pregnant og lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2003-02; Study Completion 2006-05

PRIMARY OUTCOMES:
Number of patients in remission in the two groups at the end of the treatment period

SECONDARY OUTCOMES:
Difference in time to relapse in the two treatment groups
Number of patients successfully obtaining remission
Time to remission in the two groups
Time ro relapse after study treatment is discontinued

CONTACTS AND LOCATIONS:
Overall Officials: Lone G Klinge, MD, Principal Investigator — Odense University Hospital; Jens Kjeldsen, MD, PhD, Principal Investigator — Odense University Hospital; Karsten Lauritsen, MD, Dr.med., Study Chair — Odense University Hospital; Lisbeth Ambrosius, MD,Dr.med., Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Dept. of Medical Gastroenterology (afd.S), Odense University Hospital, Odense